CLINICAL TRIAL: NCT06031428
Title: MANAGe-DM: Novel Nurse Case Management to Improve Diabetes Outcomes in Formerly Incarcerated Black Men
Acronym: MANAGe-DM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Laura Hawks, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00044942
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): All participants in the study will receive diabetes education mailers. This includes monthly mailings of diabetes education, based off the American Diabetes Association guidelines for Diabetes Education.
  Interventions: Behavioral: Monthly Educational Mailing
- MANAGe-DM (Experimental): Participants assigned to MANAGe-DM will receive the standard diabetes education mailing in addition to a novel nurse case management intervention. MANAGe-DM will include NCM services tailored to the health needs of Black men with recent release from incarceration and T2DM. MANAGe-DM will include three components: 1) diabetes education and skills training; 2) healthcare navigation and 3) basic needs navigation. . Each month of the study period, the NCM will conduct two phone call intervention sessions with individual participants.
  Interventions: Behavioral: MANAGe-DM - novel nurse case management

INTERVENTIONS:
Behavioral: MANAGe-DM - novel nurse case management — Participants assigned to MANAGe-DM will receive the standard diabetes education mailing in addition to a novel nurse case management intervention. Each month of the study period, the NCM will conduct two phone call intervention sessions with individual participants.
  Arms: MANAGe-DM
Behavioral: Monthly Educational Mailing — All participants in the study will receive diabetes education mailers. This includes monthly mailings of diabetes education, based off the American Diabetes Association guidelines for Diabetes Education. Topics covered will include diabetes basics, monitoring and medications, healthy eating and exercise, overview of common comorbidities, basics of foot care, and strategies for overcoming common pitfalls.
  Arms: Control

SUMMARY:
The study is a randomized control trial involving 100 participants (formerly incarcerated Black men with poorly controlled diabetes) to examine the effect of a tailored nurse case manager on glycemic control and other clinical outcomes, self-care behaviors, and quality of life at 6 months post-randomization.

DETAILED DESCRIPTION:
The study is a randomized control trial involving 100 participants (formerly incarcerated Black men with poorly controlled diabetes) to examine the effect of a tailored nurse case manager on glycemic control and other clinical outcomes, self-care behaviors, and quality of life at 6 months post-randomization. Participants assigned to MANAGe-DM will receive the standard diabetes education mailing in addition to a novel nurse case management intervention. Nurse case managers are trained RNs who support patients with T2DM by coordinating services, supporting self-care and implementing disease management strategies (Welch 2010). MANAGe-DM will include NCM services tailored to the health needs of Black men with recent release from incarceration and T2DM. MANAGe-DM will include three components: 1) diabetes education and skills training; 2) healthcare navigation and 3) basic needs navigation. The NCM will serve as an adjunct to the participant's primary care provider; they will not be embedded within a clinic but instead interact with the participant over the phone after study recruitment from a community setting.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* identify as Black or African American
* identify as male
* formerly incarcerated in a state or federal prison system or county jail
* clinical diagnosis of type 2 diabetes with HbA1c ≥8% at the screening visit
* able to communicate in English.

Exclusion Criteria:

* mental confusion on screening interview suggesting significant dementia
* current participation in other diabetes clinical trials
* active psychosis or acute mental disorder
* life expectancy <12 months
* awaiting arraignment, trial, sentencing in the criminal legal system
* on active surveillance by the criminal legal system, meaning on house arrest or subject to electronic monitoring

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on self-representation of gender identity
Enrollment: 100 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C | 6 months post-randomization
  Venous draw will be use to obtain HbA1C

SECONDARY OUTCOMES:
Blood Pressure | 6 months post-randomization
  Blood pressure readings (both systolic and diastolic) will be obtained using automated BP monitors programmed to take 3 readings at 2 minute intervals and give average of the 3 readings
Quality of Life (Short Form Health Survey, SF-12) | 6 months post-randomization
  The Short Form Health Survey (SF-12) version 1, developed by Ware et al. in 1996 is a valid and reliable instrument that will be used to measure quality of life. Scores will be reported in physical health related (PCS) and mental health related (MCS). Scores range from 0 to 100 with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hawks, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Center for Advancing Population Science, Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No